CLINICAL TRIAL: NCT07196839
Title: Determining the Association of TTR Stabilizing Therapy With Circulating TTR Amyloid Aggregates Over Time in Patients With ATTR-CM: Longitudinal Biomarker Study
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Justin Grodin, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-1119
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin (TTR) Amyloid Cardiomyopathy
Keywords: transthyretin; tafamidis; acoramidis; amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma and serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taking on-label TTR stabilizing treatment: Taking on-label TTR stabilizing treatment for >14 days prior to enrollment
- Initiating on-label TTR stabilizing treatment: Initiating on-label TTR stabilizing treatment within 5 days after enrollment

SUMMARY:
The objective of this study is to determine the association of clinically prescribed, on-label, TTR stabilizing therapy (e.g. tafamidis or acoramidis) with levels of circulating transthyretin amyloid aggregates (TAAs, a surrogate for amyloid disease activity) measured serially over time in patients with transthyretin cardiac amyloidosis (ATTR-CA). To accomplish this objective, the hypothesis that TTR stabilizing therapy will be associated lower circulating TAAs over time will be tested. Completion of this study will advance the understanding of the influence of ATTR-CA treatments on circulating evidence of amyloidosis and justify the role of blood testing to monitor treatment response in patients with ATTR-CA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 30-80 who have symptomatic ATTR-CA as determined by a history of HF (this will be assessed by study personnel and defined as : 1) history of hospitalization within the previous 12 months for management of HF; 2) an elevated B-type natriuretic peptide level ≥100 pg/mL or NT-proBNP ≥360 pg/mL within the previous 12 months; or 3) a clinical diagnosis of HF from a treating clinician)
* ATTR-CA previously diagnosed histologically by amyloid staining and tissue typing with immunohistochemistry or mass spectrometry or by bone scintigraphy in without abnormal M-protein
* TTR gene sequencing confirming the TTR genotype has resulted or is pending
* Enrollment will be stratified by n/N=30/50 starting on-label TTR-stabilizing therapy (e.g. tafamidis) within 5 days after enrollment or by n/N=20/50 of those currently taking TTR-stabilizing therapy

Exclusion Criteria:

* Other known causes of cardiomyopathy
* History of light-chain cardiac amyloidosis
* Cardiac transplantation
* Liver transplantation
* Has taken patisiran in the past 90 days, or inotersen in the past 180 days, has ever taken vutrisiran, or is participating in a clinical trial for ATTR treatments
* Estimated glomerular filtration rate ≤30 mL/min/1.73 m2
* Anticipated gaps in ATTR-CA treatment for 3 months after enrollment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ATTR-CA patients with a diagnosis of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Serial blood levels of circulating TTR amyloid aggregates (TAAs) | Baseline, 1 month (+/- 5 days), and 3 months (+/- 5 days).
  The primary hypothesis is that TTR stabilizing therapy will lower circulating evidence of amyloidosis in patients with ATTR-CA from baseline to 3 months. In addition, the study team expects that there will be a time*treatment interaction identifying that treatment initiation will have a differential effect on serial levels of circulating s over time than those currently on treatment. These observations will support the role for measuring circulating TAAs to monitor treatment response in ATTR-CA.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Grodin, MD MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pedretti R, Wang L, Hanna M, Benson MD, Grodin JL, Tang WHW, Masri A, Saelices L. Detection of Circulating Transthyretin Amyloid Aggregates in Plasma: A Novel Biomarker for Transthyretin Amyloidosis. Circulation. 2024 May 21;149(21):1696-1699. doi: 10.1161/CIRCULATIONAHA.123.067225. Epub 2024 May 20. No abstract available. PMID 38768274